CLINICAL TRIAL: NCT02902952
Title: Physical Exercise to Reduce Anxiety in Underserved Children With Autism Spectrum Disorders
Brief Title: Physical Exercise to Reduce Anxiety in Underserved Children With ASD
Acronym: PETRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Massachusetts General Hospital (Other); University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Jean Gehricke, Associate Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS 2016-2859
Record Dates: First submitted 2016-09-08; First posted 2016-09-16 (Estimated); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Physical Exercise Condition; Control Condition
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physical Exercise Condition (Experimental): An eight week physical exercise intervention
  Interventions: Behavioral: Physical Exercise
- Control Condition (Active Comparator): An eight week control condition consisting of sedentary activities
  Interventions: Behavioral: Control Intervention

INTERVENTIONS:
Behavioral: Physical Exercise — An eight week physical exercise intervention
  Arms: Physical Exercise Condition
Behavioral: Control Intervention — An eight week sedentary control intervention
  Arms: Control Condition

SUMMARY:
Anxiety is one of the most frequent comorbidities in children with ASD leading to poor clinical outcomes. Physical exercise has been shown to be a promising and easy to implement intervention for reducing anxiety. However, little is known about the feasibility and efficacy of physical exercise to reduce anxiety in children with ASD from underserved, low-income families. Children with ASD, ages 6 - 12 years old from low-income and Latino families will be recruited for the study and assigned to an exercise intervention group and a sedentary control group. The physical exercise program is an eight-week program, administered three times per week in small groups. Compliance, parent-rated anxiety, and salivary cortisol will be measured before and after completion of the exercise and control group interventions.

ELIGIBILITY:
Inclusion Criteria:

* Autism Spectrum Disorder (ASD) Diagnosis 6-12 years old
* ≥ 93rd percentile on CBCL or total score of ≥ 25 on SCARED
* Able to attend 3x/week for 8 consecutive weeks
* Able to follow instructions
* CalOptima Insurance or Medicaid and ability to participate in moderate physical exercise

Exclusion Criteria:

* Danger to themselves or others
* Medical conditions that may pose a risk during exercise
* Unable to participate in moderate physical exercise
* Joining a regular physical exercise program in the last 4 weeks or planning to start or discontinue a regular physical exercise program in the next 8 weeks
* Unable to attend 3x/week for 8 consecutive weeks
* Visual, auditory or motor impairments, which would preclude participation in study activities

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 148 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Anxiety rating | Change from baseline at Week 8
  Anxiety rating on the Child Behavior Checklist

SECONDARY OUTCOMES:
Salivary Cortisol | Change from baseline at Week 8
  Physiological parameter

CONTACTS AND LOCATIONS:
Overall Officials: Jean Gehricke, Ph.D., Study Chair — University of California, Irvine; Lea Ann Lowery, OTD/OTR-L, Principal Investigator — University of Missouri-Columbia
Locations (2):
- United States (2):
  - 2500 Red Hill Avenue, Santa Ana, California
  - Thompson Center for Autism, Columbia, Missouri

IPD SHARING:
Plan to Share IPD: No